CLINICAL TRIAL: NCT03369028
Title: Fitting of Commonly Available Face Masks for Late Preterm and Term Infants
Acronym: CAFF
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: CAFF
Record Dates: First submitted 2017-11-24; First posted 2017-12-11 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2017-11

CONDITIONS: Face; Newborn; Preterm Infant
MeSH Terms: conditions — Facies; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — two-dimensional and three-dimensional images retained, with no potential for DNA extraction from any retained samples. Not working with any part of the body of the investigators´ participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2d and 3D image: A 2D and 3D image of the participants' face will be taken. It will at least last 2-3 sec.
  Interventions: Other: 2D and 3D image of infants´ faces

INTERVENTIONS:
Other: 2D and 3D image of infants´ faces — 2D and 3D image of infants´ faces

SUMMARY:
Around ten percent of newborn infants require positive pressure ventilation (PPV) in the delivery room. This is most commonly delivered using a round or anatomically shaped face mask attached to a T-piece device, self-inflating bag or flow-inflating bag. Face mask ventilation is a challenging technique and difficult to ensure that an appropriate tidal volume is delivered because large and variable leaks occur between the mask and face.

It is recommended by International Guidelines to start with mask ventilation by placing a fitting face mask on the babies face.

A fitting face mask covers the mouth and nose. A non-fitting overlaps the eyes and the chin, which causes a airleak. Studies report variable leak, sometimes more than 50% of inspiratory volume, during PPV in preterm infants in the delivery room. The presence of a large leak may lead to ineffective ventilation and an unsuccessful resuscitation.

A study performed in preterm infants showed that most masks available are too big for the majority of those infants.

The investigators hypothesis is that the commonly available face masks for term infants are similarly too big for some term and late preterm infants (≥ 34 weeks gestation).

DETAILED DESCRIPTION:
The investigators would like to measure the dimensions of the faces of late preterm and term infants (≥ 34 SSW) within the first 72 hours of life and compare this data with the size of the most recommended available face masks:

VBM Germany:

external diameter smaller mask: 50 mm, external diameter bigger mask: 70 m

Laerdal:

external diameter smaller mask: 50 mm; external diameter bigger mask: 60 mm

Fisher&Paykel:

external diameter smaller mask: 50 mm; external diameter bigger mask: 60 mm

Therefore the investigators want to collect the following information from the participants:

Picture of the participant´s face (2D and 3D-Image) birth weight, head circumference, mode of delivery, gestational age, singletons/ twins/ triplets, date of birth

ELIGIBILITY:
Inclusion Criteria:

* Late preterm and term infants, gestational week ≥ 34 +0
* born at the University Hospital of Tuebingen
* signed declaration of consent from the parents
* ≤ 72 hours

Exclusion Criteria:

* congenital facial anomalies
* any respirators or other medical device that covers the face
* missing declaration of consent from the parents

Max Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Late preterm and term infants, gestational week ≥ 34 +0
  * 10 to 15 patients in every gestational-week
  * born at the University Hospital of Tuebingen
  * signed declaration of consent from the parents
  * ≤ 72 hours
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Mouth: Find out the best fitting facemask | 1 year
  Measure distance in millimeters with ImageJ and 3DMaxSoftware from the nasofrontal groove to the mental protuberance and determine if the commonly available face masks fit this study population.
Lips: Find out the best fitting facemask | 1 year
  Measure the lateral points located at each labial commissure in millimeters with ImageJ and 3DMaxSoftware and determine if the commonly available face masks fit this study population.
Eyes: Find out the best fitting facemask | 1 year
  Measure the points at the inner commissure of the eye fissure in millimeters with ImageJ and 3DMaxSoftware and determine if the commonly available face masks fit this study population.
Chin: Find out the best fitting facemask | 1 year
  Measure length of the chin in millimeters with ImageJ and 3DMaxSoftware and determine if the commonly available face masks fit this study population.

SECONDARY OUTCOMES:
Gestational age | 1 year
  Correlation between gestational age and distance from the nasofrontal groove to the mental protuberance measured in millimeters with ImageJ and 3DMaxSoftware.
Birth weight | 1 year
  Correlation between birthweight and distance from the nasofrontal groove to the mental protuberance measured in millimeters with ImageJ and 3DMaxSoftware.
headcircumference | 1 year
  Correlation between headcircumference and distance from the nasofrontal groove to the mental protuberance measured in millimeters with ImageJ and 3DMaxSoftware.
gender: male/female | 1 year
  Correlation between gender (male/female) and distance from the nasofrontal groove to the mental protuberance measured in millimeters with ImageJ and 3DMaxSoftware.
way of delivery: spontaneous/cesarean | 1 year
  Correlation between way of delivery and distance from the nasofrontal groove to the mental protuberance measured in millimeters with ImageJ and 3DMaxSoftware..

CONTACTS AND LOCATIONS:
Locations (1):
- University clinic tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sawyer T, Umoren RA, Gray MM. Neonatal resuscitation: advances in training and practice. Adv Med Educ Pract. 2016 Dec 23;8:11-19. doi: 10.2147/AMEP.S109099. eCollection 2017. PMID 28096704
- [Background] Singhal N, McMillan DD, Yee WH, Akierman AR, Yee YJ. Evaluation of the effectiveness of the standardized neonatal resuscitation program. J Perinatol. 2001 Sep;21(6):388-92. doi: 10.1038/sj.jp.7210551. PMID 11593374
- [Background] Wyllie J, Bruinenberg J, Roehr CC, Rudiger M, Trevisanuto D, Urlesberger B. European Resuscitation Council Guidelines for Resuscitation 2015: Section 7. Resuscitation and support of transition of babies at birth. Resuscitation. 2015 Oct;95:249-63. doi: 10.1016/j.resuscitation.2015.07.029. Epub 2015 Oct 15. No abstract available. PMID 26477415
- [Background] O'Donnell CP, Davis PG, Morley CJ. Positive pressure ventilation at neonatal resuscitation: review of equipment and international survey of practice. Acta Paediatr. 2004 May;93(5):583-8. doi: 10.1111/j.1651-2227.2004.tb02981.x. PMID 15174776
- [Background] O'Donnell CP, Davis PG, Lau R, Dargaville PA, Doyle LW, Morley CJ. Neonatal resuscitation 2: an evaluation of manual ventilation devices and face masks. Arch Dis Child Fetal Neonatal Ed. 2005 Sep;90(5):F392-6. doi: 10.1136/adc.2004.064691. Epub 2005 May 4. PMID 15871989
- [Background] Schmolzer GM, Kamlin OC, O'Donnell CP, Dawson JA, Morley CJ, Davis PG. Assessment of tidal volume and gas leak during mask ventilation of preterm infants in the delivery room. Arch Dis Child Fetal Neonatal Ed. 2010 Nov;95(6):F393-7. doi: 10.1136/adc.2009.174003. Epub 2010 Jun 14. PMID 20547584
- [Background] Cheung D, Mian Q, Cheung PY, O'Reilly M, Aziz K, van Os S, Pichler G, Schmolzer GM. Mask ventilation with two different face masks in the delivery room for preterm infants: a randomized controlled trial. J Perinatol. 2015 Jul;35(7):464-8. doi: 10.1038/jp.2015.8. Epub 2015 Feb 26. PMID 25719544
- [Background] Kumar VH, Skrobacz A, Ma C. Impact of bradycardia or asystole on neonatal cardiopulmonary resuscitation at birth. Pediatr Int. 2017 Aug;59(8):891-897. doi: 10.1111/ped.13310. Epub 2017 Jul 9. PMID 28452098
- [Background] Wood FE, Morley CJ, Dawson JA, Kamlin CO, Owen LS, Donath S, Davis PG. Improved techniques reduce face mask leak during simulated neonatal resuscitation: study 2. Arch Dis Child Fetal Neonatal Ed. 2008 May;93(3):F230-4. doi: 10.1136/adc.2007.117788. Epub 2007 Nov 26. PMID 18039750
- [Background] Wood FE, Morley CJ. Face mask ventilation--the dos and don'ts. Semin Fetal Neonatal Med. 2013 Dec;18(6):344-51. doi: 10.1016/j.siny.2013.08.009. Epub 2013 Sep 14. PMID 24041823
- [Background] Finer NN, Rich W, Wang C, Leone T. Airway obstruction during mask ventilation of very low birth weight infants during neonatal resuscitation. Pediatrics. 2009 Mar;123(3):865-9. doi: 10.1542/peds.2008-0560. PMID 19255015
- [Background] Deindl P, Schwindt J, Berger A, Schmolzer GM. An instructional video enhanced bag-mask ventilation quality during simulated newborn resuscitation. Acta Paediatr. 2015 Jan;104(1):e20-6. doi: 10.1111/apa.12826. Epub 2014 Oct 30. PMID 25308155
- [Background] O'Shea JE, Thio M, Owen LS, Wong C, Dawson JA, Davis PG. Measurements from preterm infants to guide face mask size. Arch Dis Child Fetal Neonatal Ed. 2016 Jul;101(4):F294-8. doi: 10.1136/archdischild-2014-307350. Epub 2015 Apr 10. PMID 25862726
- [Background] Krimmel M, Kluba S, Breidt M, Bacher M, Dietz K, Buelthoff H, Reinert S. Three-dimensional assessment of facial development in children with Pierre Robin sequence. J Craniofac Surg. 2009 Nov;20(6):2055-60. doi: 10.1097/SCS.0b013e3181be87db. PMID 19881369
- [Background] Krimmel M, Kluba S, Breidt M, Bacher M, Muller-Hagedorn S, Dietz K, Bulthoff H, Reinert S. Three-dimensional assessment of facial development in children with unilateral cleft lip with and without alveolar cleft. J Craniofac Surg. 2013 Jan;24(1):313-6. doi: 10.1097/SCS.0b013e318275ed60. PMID 23348308
- [Background] Farkas LG. Accuracy of anthropometric measurements: past, present, and future. Cleft Palate Craniofac J. 1996 Jan;33(1):10-8; discussion 19-22. doi: 10.1597/1545-1569_1996_033_0010_aoampp_2.3.co_2. PMID 8849854
- [Background] Schneider CA, Rasband WS, Eliceiri KW. NIH Image to ImageJ: 25 years of image analysis. Nat Methods. 2012 Jul;9(7):671-5. doi: 10.1038/nmeth.2089. PMID 22930834
- [Background] Farkas LG. [Centenary of Ambrus Abraham]. Orv Hetil. 1994 Jun 26;135(26):1429. No abstract available. Hungarian. PMID 8028900
- [Derived] Haase B, Badinska AM, Maiwald CA, Poets CF, Springer L. Comparison of nostril sizes of newborn infants with outer diameter of endotracheal tubes. BMC Pediatr. 2021 Sep 23;21(1):417. doi: 10.1186/s12887-021-02889-5. PMID 34556062
- [Derived] Haase B, Badinska AM, Koos B, Poets CF, Lorenz L. Do commonly available round facemasks fit near-term and term infants? Arch Dis Child Fetal Neonatal Ed. 2020 Jul;105(4):364-368. doi: 10.1136/archdischild-2019-317531. Epub 2019 Sep 21. PMID 31542729